CLINICAL TRIAL: NCT03752931
Title: Prevention of Postoperative Cardiac Arrythmias in Thoracic Surgery : Celiprolol Versus Diltiazem
Brief Title: Celiprolol Versus Ditiazem for the Prevention of Postoperative Cardiac Arrythmias in Thoracic Surgery
Acronym: CelDilPreCA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abderrahmane Mami Hospital (Other)
Responsible Party: Principal Investigator, MahmoudMARZOUK, Medical Doctor anesthesiology and intensive care, Abderrahmane Mami Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: MAMICELDIL
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Cardiac Complication
Keywords: Pneumonectomy Thoracic surgery Celiprolol Diltiazem
MeSH Terms: interventions — Celiprolol; Diltiazem

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Celiprolol (Active Comparator): receiving 1 tablet per day of celiprolol (Celiprol®) 200 mg in the morning from the first postoperative day after pneumonectomy or bi lobecomty for 2 weeks.
  Interventions: Drug: Celiprolol
- Diltiazem (Active Comparator): receiving 1 capsule per day of diltiazem (Monotildiem® LP) 200 mg in the morning from the first postoperative day after pneumonectomy or bi lobectomy for 2 weeks.
  Interventions: Drug: Diltiazem

INTERVENTIONS:
Drug: Celiprolol — receiving 1 tablet per day of Celiprolol 200 mg in the morning from the first postoperative day after pneumonectomy or bi lobecomty for 2 weeks.
  Arms: Celiprolol
Drug: Diltiazem — receiving 1 tablet per day of Diltiazem 200 mg in the morning from the first postoperative day after pneumonectomy or bi lobecomty for 2 weeks.
  Arms: Diltiazem

SUMMARY:
Cardiac arrythmias are the most common cardiac complications after thoracic surgery. They are made primarily of postoperative atrial fibrillation (POAF).

They are associated with an increased risk of stroke, increased length of hospital stay and cost of care, and increased long-term mortality.

Randomized , single-blind prospective study in the anesthesia and intensive care department of Abderrahmen Mami hospital Ariana Tunisia comparing the efficacy of Diltiazem versus Celiprolol in the prevention of postoperative cardiac arrythmias in patients proposed for pneumonectomy and bilobectomy.

DETAILED DESCRIPTION:
Cardiac arrythmias are the most common cardiac complications after thoracic surgery. They are made primarily of postoperative atrial fibrillation (POAF).

They are associated with an increased risk of stroke, increased length of hospital stay and cost of care, and increased long-term mortality.

According to the American Association of Thoracic Surgery (AATS), interventions at high risk for FAPO (> 15%) are: anterior mediastinal mass resection, thoracoscopic lobectomy, thoracotomy lobectomy, pneumonectomy, pleurectomy, tracheal resection, emphysema bubble, bronchopleural fistula repair, lung transplantation and oesophagectomy. And it has been shown that the occurrence of postoperative atrial fibrillation is correlated with the extent of resection in case of lung resection surgery such as lobectomy or pneumonectomy.

Based on their multifactorial etiology, different pharmacological classes have been used for the prevention of POAF with varying degrees of success such as Amiodarone, Digoxin, Flecaine, Magnesium Sulfate, Beta Blockers, Calcium Inhibitors and Statins.

Recommendations were made for the prevention of POAF by the Society of Thoracic Surgeons (STS) in 2011 and the AATS in 2014 and concluded that Diltiazem is recommended for prevention and it is a Grade IIA for recommendations of 2011 and a grade IIB for the 2014 recommendations. Beta-blockers (BB) are recommended and it is a grade IIB for the 2011 recommendations. In addition, amiodarone is not recommended in case of pneumonectomy because of of its pulmonary toxicity for the 2011 recommendations and is ranked grade IIA for the 2014 recommendations.

A meta-analysis published in Chest in 2017 involving 22 studies and 2891 patients showed that the pharmacological prevention of postoperative rhythm disorders after thoracic surgery decreases their incidence but does not reduce mortality in the short term. Several drugs have been studied. Betablockers have the probability of being the most effective agent. Calcium inhibitors are less effective.

In view of these conflicting results and in the absence of a large randomized controlled trial comparing two pharmacologic agents for the prevention of POAF, a certain degree of uncertainty persists regarding the superiority of one agent over another. especially in case of pulmonary resection surgery. Most studies compare drugs versus placebo. Among these drugs Diltiazem and BB are among the most effective and safe.

Randomized , single-blind prospective study in the anesthesia and chest surgery departments of Abderrahmen Mami hospital Ariana Tunisia.

The objective is to compare the efficacy of Celiprolol -Class II of cardioselective anti-arrhythmic B1 with B2 agonist activity with intrinsic sympathomimetic activity- versus Diltiazem -Class IV antiarrhythmic calcium antagonist with direct cardiac effects- in the prevention of cardiac arrhythmias after thoracic surgery such as bilobectomy and pneumonectomy.

Have been included:

* Age ≥ 18 years
* Sinus rhythm preoperatively.
* Surgery at high risk of atrial arrhythmia occurring postoperatively:

Bi-lobectomy Pneumonectomy

Have not been included:

* history of cardiac arrhythmia.
* A prior history of atrio-ventricular block with non-paired degrees II or III.
* Patients on calcium channel blockers or beta-blockers as background therapy.
* Hypersensitivity to Diltiazem and / or Celiprolol and / or any of the excipients.
* Renal insufficiency with creatinine clearance <40 ml / min.
* wolf parkinson white syndrome.
* Myasthenia gravis.
* Chronic Obstructive Pulmonary Disease: GOLD III or IV.

Have been excluded :

• Signs of myocardial ischemia per or post operative.

• Persistent postoperative hypotension requiring the use of catecholamines.

* Persistent bradycardia.
* Decompensated cardiac insufficiency.
* Acute bowel obstruction.

  * The main criterion of judgment:
* Incidence of early postoperative atrial fibrillation.

  * Secondary criteria for judgment:
* The incidence of late arrhythmia (> 14 days) during or after hospitalization during the 30 postoperative days.
* The incidence of other rhythm disorders.
* The duration of the arrhythmia in case of occurrence.
* Length of stay in intensive care unit and hospital.
* 30-day mortality.
* Other complications during 14 days postoperative:

Pulmonary: Atelectasis, pneumonitis, ARDS, Cardiovascular: heart failure, heart attack, pulmonary embolism. Neurological: stroke Acute renal failure. • Product Tolerance: Digestive Disorders, Dizziness, Bradycardia, Hypotension, Bronchospasm, Hypoglycemia or Hyperglycemia.

* Perioperative management:

- Preoperatively:

All patients are assessed at the pre-anesthetic consultation. All patients are informed about postoperative treatment to reduce the incidence of arrhythmias.

A consent form is signed for this purpose.

* Inoperative:
* General anaesthesia:

Induction: Fentanyl, Propofol, Cisatracurium Maintenance: Propofol to push electric syringe, fentanyl and cisatracurium.

* Perioperative fluid restriction <25ml / kg / 24h with isotonic saline as much as possible.
* The extent of pericardial resection and mediastinal lymph node dissection are mentioned.
* Bleeding estimated peroperatively, the need for catecholamines, labile blood products and intraoperative incidents are noted.
* Postoperative analgesia combines Paracetamol 1g per 6 hours with thoracic epidural analgesia or multimodal analgesia with morphine titration as needed.

Postoperatively:

- All patients are admitted to intensive care.

* Close monitoring of hemodynamic, respiratory and neurological parameters.
* Patients are randomized into 2 groups:

Group 1: receiving 1 tablet per day of celiprolol 200 mg in the morning from the first day after surgery.

Group 2: receiving 1 capsule per day of diltiazem 200 mg in the morning from the first postoperative day.

The target heart rate is between 70 and 80 bpm by titrating the antiarrhythmic agent.

The treatment will be continued for 14 days.

* electrocardiogram at 6 hours postoperative or if clinical suspicion of arrhythmia or modification to the scope then twice a day.
* Postoperative blood count.
* Magnesemia, phosphoremia, calcemia, and blood ionogram at the first postoperative day and correction if abnormalities.
* X-ray of the postoperative chest and 1 time per day especially for the research of deviation of the mediastinum in case of pneumonectomy.

The occurrence of an arrhythmia will be treated according to the following algorithm:

* Look for probable cause of bleeding, pulmonary embolism, pneumothorax, pericardial effusion, mediastinal deviation, hypoxia, myocardial ischemia or sepsis.
* Optimize the volemia.
* Correct metabolic disorders.
* Optimize analgesia.
* If hemodynamically unstable:

Of duration <48 h: external electric shock and advice cardiology. Duration> 48 h: consider anticoagulation, external electrical shock and cardiology.

-It is hemodynamically stable

Duration <48h:

Consider anticoagulation if CHA2DS2 score VASc> 1, amiodarone IV then per os and notice cardiology.

Duration> 48h: consider anticoagulation, IV amiodarone then per os and opinion cardiology.

• All patients are referred to outpatient cardiology consultations with a rhythmic holter upon discharge.

The occurrence of another postoperative complication will be noted by specifying the date of occurrence in relation to the arrhythmia:

* Pulmonary: Atelectasis, pneumonitis, ARDS, need for prolonged mechanical ventilation.
* Cardiovascular: heart failure, myocardial infarction, pulmonary embolism.
* Neurological: Stroke
* Acute renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years Sinus rhythm preoperatively.

Surgery at high risk of atrial arrhythmia occurring postoperatively:

* Bi-lobectomy
* Pneumonectomie

Exclusion Criteria:

* Signs of myocardial ischemia per or post operative.
* Persistent postoperative hypotension requiring the use of catecholamines.
* Persistent bradycardia
* Decompensated cardiac insufficiency.
* Acute intestinal obstruction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
incidence of early postoperative atrial fibrillation | 14 days

SECONDARY OUTCOMES:
incidence of other cardiac arrythmias and other complications | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marzouk Mahmoud, MD, Principal Investigator — Abderrahmane Mami Hospital
Locations (1):
- Hospital Abderrahmane Mami, Aryanah, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao BC, Huang TY, Deng QW, Liu WF, Liu J, Deng WT, Liu KX, Li C. Prophylaxis Against Atrial Fibrillation After General Thoracic Surgery: Trial Sequential Analysis and Network Meta-Analysis. Chest. 2017 Jan;151(1):149-159. doi: 10.1016/j.chest.2016.08.1476. Epub 2016 Oct 8. PMID 27729264
- [Background] Fernando HC, Jaklitsch MT, Walsh GL, Tisdale JE, Bridges CD, Mitchell JD, Shrager JB. The Society of Thoracic Surgeons practice guideline on the prophylaxis and management of atrial fibrillation associated with general thoracic surgery: executive summary. Ann Thorac Surg. 2011 Sep;92(3):1144-52. doi: 10.1016/j.athoracsur.2011.06.104. No abstract available. PMID 21871327
- [Background] Frendl G, Sodickson AC, Chung MK, Waldo AL, Gersh BJ, Tisdale JE, Calkins H, Aranki S, Kaneko T, Cassivi S, Smith SC Jr, Darbar D, Wee JO, Waddell TK, Amar D, Adler D; American Association for Thoracic Surgery. 2014 AATS guidelines for the prevention and management of perioperative atrial fibrillation and flutter for thoracic surgical procedures. J Thorac Cardiovasc Surg. 2014 Sep;148(3):e153-93. doi: 10.1016/j.jtcvs.2014.06.036. Epub 2014 Jun 30. No abstract available. PMID 25129609